CLINICAL TRIAL: NCT07069049
Title: Electroacupuncture in the Treatment of Patients Undergoing Transperineal Prostate Biopsy Under Local Anesthesia: a Randomized, Single-blind, Sham-electroacupuncture Parallel Control, Multi-center Clinical Trial
Brief Title: Electroacupuncture in the Treatment of Patients Undergoing Transperineal Prostate Biopsy Under Local Anesthesia
Acronym: EATPULA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiangyang Zhan, Physician in Charge, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1592-175-01
Record Dates: First submitted 2025-05-20; First posted 2025-07-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: electroacupuncture; Prostate Needle biopsy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupunture (Experimental): In the EA group, on the basis of routine local lidocaine anesthesia, EA stimulation was performed 20min before the operation and the needles were retained until the completion of the operation. Sterile acupuncture needles (Huatuo brand, specification: 0.25mm*40mm) were applied to Hegu (Li4), Neiguan (PC 6), Guanyuan (CV 4) and Sanyinjiao (SP 6) by twidling, rotating, lifting and thrusting for 30 seconds. After getting qi (a feeling of acid, numbness, weight and swelling), the electronic acupuncture instrument (SDZ-II type, Huatuo brand) was connected, and the continuous wave was 50HZ. The current intensity was 1-5mA (preferably as much as the patient could tolerate without pain). Acupuncture was performed by a fixed-practice acupuncturist with at least 5 years of experience. Acupuncturists were trained in acupoints and acupuncture manipulation before the trial, and intervention completion was recorded.
  Interventions: Other: electroacupuncture
- Sham-electroacupunture (Sham Comparator): The intervention process of patients in the control group was the same as that of the experimental group, but the acupuncture site was located 3mm away from the acupoints of the experimental group, and the acupuncture method was shallow acupuncture, only 1-4mm through the skin. After the sham acupuncture, the lifting and thrusting twisling method was not performed to avoid qi gain. The needles were removed if the patient experienced any adverse events related to acupuncture. Sham acupuncture was performed by a fixed-practice acupuncturist with at least 5 years of experience. Acupuncturists were trained in sham acupoints and acupuncture manipulation before the trial, and intervention completion was recorded.
  Interventions: Other: Sham-electroacupunture

INTERVENTIONS:
Other: electroacupuncture — Sterile acupuncture needles (Huatuo brand, specification: 0.25mm*40mm) were applied to Hegu (Li4), Neiguan (PC 6), Guanyuan (CV 4) and Sanyinjiao (SP 6) by twidling, rotating, lifting and thrusting for 30 seconds. After getting qi (a feeling of acid, numbness, weight and swelling), the electronic acupuncture instrument (SDZ-II type, Huatuo brand) was connected, and the continuous wave was 50HZ. The current intensity was 1-5mA (preferably as much as the patient could tolerate without pain).
  Arms: electroacupunture
Other: Sham-electroacupunture — Sham electroacupuncture was applied at the non-meridian and non-acupoint sites 3mm apart from the acupoints in the experimental group. The acupuncture method was shallow acupuncture, only 1-4mm through the skin.
  Arms: Sham-electroacupunture

SUMMARY:
Prostate biopsy is the gold standard for the diagnosis of prostate cancer, and transperineal puncture is a common approach. It has the advantages of no bowel preparation and relative safety. At present, transperineal puncture is often performed under local anesthesia, but there are still clinical problems such as pain and anxiety for patients. Electroacupuncture is often used as an auxiliary means of local anesthesia in China, which has the advantages of analgesia and anti-anxiety. This study was conducted to evaluate the efficacy and safety of electroacupuncture combined with local anesthesia in transperineal needle biopsy.

DETAILED DESCRIPTION:
Prostate cancer ranks the first in the incidence of male malignant tumors and the second in mortality in the world, which seriously affects men's physical and mental health. At present, the gold standard for the diagnosis of prostate cancer is prostate biopsy. Transrectal biopsy and transperineal biopsy are commonly used. There is no significant difference in the detection rate of prostate cancer between the two methods, but each has its advantages and disadvantages. Transrectal prostate biopsy can be performed with local anesthesia, but the risk of postoperative infection is high. After transrectal prostate biopsy, bacteriuria was detected in 44% of patients and bacteremia in 16%, with infection as the leading cause of rehospitalization within 2 weeks after discharge (81%). Transperineal prostate biopsy does not require bowel preparation, and the risk of infection is minimal. However, this approach is prone to significant pain, and most cases are completed by general anesthesia. However, the operation time of general anesthesia is long, the economic cost is high, and the majority of prostate biopsy patients are elderly patients, with more underlying heart and lung diseases, and the risk of anesthesia is high. The convenience of local anesthesia and out-patient biopsy will be the development trend of prostate biopsy in the future. However, pain and anxiety caused by local anesthesia are not negligible factors during prostate biopsy. Studies have shown that approximately 50% of patients experience moderate or greater pain during prostate biopsy under local anesthesia. The use of analgesic drugs such as lidocaine gel and non-steroidal anti-inflammatory drugs (such as diclofenac) can not significantly reduce the pain caused by probe manipulation and biopsy sampling. In the process of local anesthesia surgery, due to the interaction between anxiety and pain for surgery, patients will also have vagal symptoms such as decreased blood pressure and bradycardia, which will increase the risk of surgery. In clinical practice, some patients give up pathological biopsy due to the fear of puncture, thus missing the best period of diagnosis and treatment. Therefore, reducing the anxiety and pain caused by prostate biopsy is the key link to complete prostate biopsy under local anesthesia.

Acupuncture and moxibustion is an important part of traditional Chinese medicine, which can be divided into hand acupuncture and electroacupuncture. Electroacupuncture is a way of stimulating acupoints by connecting appropriate current after hand acupuncture to get qi, which can enhance the sensation of acupuncture and play a continuous stimulating effect on acupoints, thus enhancing the therapeutic effect of acupuncture and moxibustion. Electroacupuncture has clinically significant effects on many types of pain management. Studies have shown that electroacupuncture has a significant effect on perioperative analgesia and can improve patients' satisfaction with surgery. In addition, electroacupuncture can also relieve perioperative anxiety, reduce stress response, and maintain the stability of cardiopulmonary function during the operation. Our previous observational study has shown that electroacupuncture can reduce the pain score and anxiety score of patients undergoing perineal prostate biopsy under local anesthesia, improve the surgical cooperation, without postoperative complications and high patient satisfaction. At present, electroacupuncture is not recommended as a analgesic and anti-anxiety regimen in prostate biopsy guidelines. In order to further verify the analgesic and anti-anxiety effect of electroacupuncture in prostate biopsy under local anesthesia, improve the level of clinical evidence, and provide a basis for clinical promotion in the future, it is necessary to conduct high-quality randomized controlled and multi-center clinical trials.

This study was a randomized, single-blind, placebo-controlled, multi-center clinical trial. After the subjects met the inclusion and exclusion criteria were included, they were randomly assigned to the electroacupuncture group and the sham electroacupuncture group according to the ratio of 1:1. The potential mechanism of EA in relieving pain and anxiety was explored.

ELIGIBILITY:
Inclusion Criteria:

- (1) To voluntarily participate in the study, I or his legal representative signed a written informed consent.

(2) 18-80 years old (including 18 and 80 years old), male. (3) in accordance with the indication of prostate biopsy.

Exclusion Criteria:

* (1) in the stage of acute genitourinary infection or fever. (2) patients with chronic pain (such as bone metastasis of prostate cancer, knee osteoarthritis, scapulohumeral periarthritis, etc.) or acute pain (tonsillitis, acute lumbar sprain, etc.) before surgery.

  (3) Continuous use of anti-anxiety or analgesic drugs (use of anti-anxiety drugs or analgesics for more than 1 week in the past 3 months).

  (4) in the decompensated stage of cardiac insufficiency; A disease with a tendency to bleed heavily.

  (5) severe immunosuppression. (6) hypertension, diabetes and other complications were poorly controlled or unstable.

  (7) complicated with severe internal or external hemorrhoids, perianal or rectal lesions, and anal stenosis.

  (8) perineal skin ulceration, infection, and abnormal skin sensation. (9) patients with serious psychological diseases or uncooperative puncture. (10) allergy to narcotic drugs and fear of acupuncture operators. (11) Participants who participated in other clinical trials within 3 months before enrollment.

  (12) other conditions considered by the investigator to be inappropriate to participate in the trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
The maximum pain level | The end of the operation
  Use Numerical Rating Scale to Assess the maximum pain level during the operation,0-100mm,higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Area under the curve for cumulative pain scores | 1h、6h、24h after completion of surgery
  Use Numerical Rating Scale to Assess the maximum pain level in 1h-24h after after the completion of surgery
Visual Analogue Scale for anxiety | At the beginning of operation and at the completion of operation
  Visual Analogue Scale for anxiety, 0-10,higher scores mean a worse outcome.
Incidence of rescue analgesia and total number of rescue analgesia | At the completion of operation
  Incidence and number
Blood pressure | At the completion of the operation and 20 min before the start of the operation
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Zhan Xiangyang, Principal Investigator — Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine